CLINICAL TRIAL: NCT01829750
Title: Phase 2 Study of Intracoronary Infusion of Cardiac Progenitor Cells in Patients With Univentricular Heart Disease
Brief Title: Cardiac Progenitor Cell Infusion to Treat Univentricular Heart Disease (PERSEUS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Okayama University (Other)
Collaborators: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Principal Investigator, Hidemasa Oh, MD, Professor, Okayama University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0329-18; MHLW25040101 (Other Grant/Funding Number: MHLW25040101)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Hypoplastic Left Heart Syndrome; Single Right Ventricle; Single Left Ventricle
Keywords: Univentricular heart
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): (Stage 1) No active intervention after standard surgical treatment
  (Stage 2) Rescuing transplantation by cardiac progenitor cell infusion is applicable in patients, along with their written consent, 4 months after palliations who were assigned as control group in stage 1.
  Interventions: Genetic: Cardiac progenitor cell infusion
- Cardiac progenitor cell infusion (Active Comparator): (Stage 1) single dose, intracoronary infusion of 0.3 million cells/kg cardiac progenitor cells
  Interventions: Genetic: Cardiac progenitor cell infusion

INTERVENTIONS:
Genetic: Cardiac progenitor cell infusion — (Stage 1) Cardiac progenitor cell infusion in patients who assigned as active comparator group
  (Stage 2) Rescuing transplantation is applicable in patients, along with their written consent, 4 months after palliations who were allocated as control group in stage 1.

SUMMARY:
The purpose of this study is to investigate the efficacy of intracoronary infusion of cardiac progenitor cells in patients with univentricular heart disease. Patients with preoperative high-risk group or whose cardiac function did not recover postoperatively eventually have no choice other than heart transplantation.

DETAILED DESCRIPTION:
Following the safety verification of the Phase I study (TICAP trial) that has been implemented and completed, the efficacy will be verified in this Phase II clinical study. The rationale of this study is based on the animal studies that transplanted cardiac progenitor cells may regenerate damaged myocardium by giving rise to cardiac muscle and vascular cell types. Preclinical and phase I studies indicate the possibilities of cardiac function improvements and reduced myocardial fibrosis by progenitor cell infusion.

The efficacy of cell transplantation is assessed as the primary endpoint of the Phase II clinical study. The improvements of cardiac ejection fraction assessed by echocardiography, ventriculography, and cardiac MRI, which are conducted before and after treatment, are assessed as the evaluation items. The absolute values of the improvement of cardiac ejection fraction obtained by the above three imaging modalities before and after treatment are compared between two groups of the transplantation group and non-transplantation group.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Age is 0 year or more and 20 years or less at the time of enrollment.
2. The patients have functional single ventricular physiology with the indication to have stage-2 or -3 palliative surgeries.
3. The ventricular ejection fraction <60%.

Exclusion Criteria:

1. Cardiogenic shock
2. A patient with unstoppable extracorporeal circulation
3. A patient with lethal, uncontrollable arrhythmia
4. A patient with a complication of coronary artery disease
5. A patient with a complication of brain dysfunction due to circulatory failure
6. A patient with malignant neoplasm
7. A patient with a complication of serious neurologic disorder
8. A patient with high-grade pulmonary embolism or pulmonary hypertension
9. A patient with high-grade renal failure
10. A patient with multiple organ failure
11. Active infection (including endocarditis)
12. Sepsis
13. Active hemorrhagic disease (e. g. gastrointestinal bleeding, injury)

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cardiac function | 3 Months
  The primary outcome measure is to evaluate the cardiac function improvement by echocardiography, ventriculography, and cardiac MRI, which are conducted before and 3 months after surgical treatment.

SECONDARY OUTCOMES:
Cardiac function | 12 Months
  The secondary outcome measure is to determine the cardiac function improvements by three different imaging modalities at 12 months after treatment.

OTHER OUTCOMES:
Clinical symptoms | 3 and 12 Months
  Clinical symptoms and BNP levels will be assessed at 3- and 12-months after treatment and compared with control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hidemasa Oh, M.D., Ph.D., Principal Investigator — Okayama University
Locations (1):
- Okayama University, Okayama, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh H, Bradfute SB, Gallardo TD, Nakamura T, Gaussin V, Mishina Y, Pocius J, Michael LH, Behringer RR, Garry DJ, Entman ML, Schneider MD. Cardiac progenitor cells from adult myocardium: homing, differentiation, and fusion after infarction. Proc Natl Acad Sci U S A. 2003 Oct 14;100(21):12313-8. doi: 10.1073/pnas.2132126100. Epub 2003 Oct 6. PMID 14530411
- [Background] Tateishi K, Ashihara E, Honsho S, Takehara N, Nomura T, Takahashi T, Ueyama T, Yamagishi M, Yaku H, Matsubara H, Oh H. Human cardiac stem cells exhibit mesenchymal features and are maintained through Akt/GSK-3beta signaling. Biochem Biophys Res Commun. 2007 Jan 19;352(3):635-41. doi: 10.1016/j.bbrc.2006.11.096. Epub 2006 Nov 27. PMID 17150190
- [Background] Tateishi K, Ashihara E, Takehara N, Nomura T, Honsho S, Nakagami T, Morikawa S, Takahashi T, Ueyama T, Matsubara H, Oh H. Clonally amplified cardiac stem cells are regulated by Sca-1 signaling for efficient cardiovascular regeneration. J Cell Sci. 2007 May 15;120(Pt 10):1791-800. doi: 10.1242/jcs.006122. PMID 17502484
- [Background] Tateishi K, Takehara N, Matsubara H, Oh H. Stemming heart failure with cardiac- or reprogrammed-stem cells. J Cell Mol Med. 2008 Dec;12(6A):2217-32. doi: 10.1111/j.1582-4934.2008.00487.x. Epub 2008 Aug 27. PMID 18754813
- [Background] Takehara N, Tsutsumi Y, Tateishi K, Ogata T, Tanaka H, Ueyama T, Takahashi T, Takamatsu T, Fukushima M, Komeda M, Yamagishi M, Yaku H, Tabata Y, Matsubara H, Oh H. Controlled delivery of basic fibroblast growth factor promotes human cardiosphere-derived cell engraftment to enhance cardiac repair for chronic myocardial infarction. J Am Coll Cardiol. 2008 Dec 2;52(23):1858-1865. doi: 10.1016/j.jacc.2008.06.052. PMID 19038683
- [Result] Ishigami S, Ohtsuki S, Eitoku T, Ousaka D, Kondo M, Kurita Y, Hirai K, Fukushima Y, Baba K, Goto T, Horio N, Kobayashi J, Kuroko Y, Kotani Y, Arai S, Iwasaki T, Sato S, Kasahara S, Sano S, Oh H. Intracoronary Cardiac Progenitor Cells in Single Ventricle Physiology: The PERSEUS (Cardiac Progenitor Cell Infusion to Treat Univentricular Heart Disease) Randomized Phase 2 Trial. Circ Res. 2017 Mar 31;120(7):1162-1173. doi: 10.1161/CIRCRESAHA.116.310253. Epub 2017 Jan 4. PMID 28052915
- [Derived] Hirai K, Sawada R, Hayashi T, Araki T, Nakagawa N, Kondo M, Yasuda K, Hirata T, Sato T, Nakatsuka Y, Yoshida M, Kasahara S, Baba K, Oh H; TICAP/PERSEUS Study Group. Eight-Year Outcomes of Cardiosphere-Derived Cells in Single Ventricle Congenital Heart Disease. J Am Heart Assoc. 2024 Nov 19;13(22):e038137. doi: 10.1161/JAHA.124.038137. Epub 2024 Nov 11. PMID 39526355
- [Derived] Sano T, Ousaka D, Goto T, Ishigami S, Hirai K, Kasahara S, Ohtsuki S, Sano S, Oh H. Impact of Cardiac Progenitor Cells on Heart Failure and Survival in Single Ventricle Congenital Heart Disease. Circ Res. 2018 Mar 30;122(7):994-1005. doi: 10.1161/CIRCRESAHA.117.312311. Epub 2018 Jan 24. PMID 29367212